CLINICAL TRIAL: NCT01308138
Title: Study of Gaining Further Understanding of the Underlying Mechanisms of Myocardial Function
Brief Title: Myocardial Physiology And Microanatomy In Individuals Undergoing Heart Surgery
Acronym: TRIMRIPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: TRIMRIPC
Record Dates: First submitted 2011-02-02; First posted 2011-03-03 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Myocardial Injury
Keywords: Physical Activity; pathology; Physical Deconditioning
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ExerciseTr (Experimental)
  Interventions: Behavioral: Exercise training
- Remote ischemic preconditioning group (Experimental)
  Interventions: Procedure: remote ischemic preconditioning
- Control patient group (No Intervention)

INTERVENTIONS:
Behavioral: Exercise training — exercise training
  Arms: ExerciseTr
Procedure: remote ischemic preconditioning — remote ischemic preconditioning
  Arms: Remote ischemic preconditioning group

SUMMARY:
The main focus of the project is to determine to what degree myocardial energy metabolism is linked to impaired function in human cardiomyocytes, whether exercise training and remote ischemic preconditioning can restore cardiomyocyte function and whether this is linked to improved mitochondrial and cell function.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary heart surgery and heart transplantation

Exclusion Criteria:

* myocardial infarction closer than 4 weeks to project start, serious valve defects, diabetes, unstable angina, uncontrolled hypertension, kidney failure (creatinin > 140)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Mitochondrial respiration | 1 hour
  Oxygraph (Strathkelvin)

CONTACTS AND LOCATIONS:
Overall Officials: Katrine Hordnes, MD, Principal Investigator — National Taiwan Normal University
Locations (1):
- Norwegian University of Science and Technology, Medical Faculty, Trondheim, Sør-Trondelag, Norway

REFERENCES:
- [Result] Slagsvold KH, Moreira JB, Rognmo O, Hoydal M, Bye A, Wisloff U, Wahba A. Remote ischemic preconditioning preserves mitochondrial function and activates pro-survival protein kinase Akt in the left ventricle during cardiac surgery: a randomized trial. Int J Cardiol. 2014 Dec 15;177(2):409-17. doi: 10.1016/j.ijcard.2014.09.206. Epub 2014 Oct 14. PMID 25456576
- [Derived] Slagsvold KH, Rognmo O, Hoydal M, Wisloff U, Wahba A. Remote ischemic preconditioning preserves mitochondrial function and influences myocardial microRNA expression in atrial myocardium during coronary bypass surgery. Circ Res. 2014 Feb 28;114(5):851-9. doi: 10.1161/CIRCRESAHA.114.302751. Epub 2013 Dec 26. PMID 24371264